CLINICAL TRIAL: NCT01421979
Title: Clinical Trial on the Effects of Caffeine and Taurine From Energy Drinks (EDs) to Parameters of the Cardiovascular System in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ED2011
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Cardiovascular Risk
MeSH Terms: interventions — Energy Drinks; Taurine; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- exposure under sleep deprivation (Experimental): Examination of the effects of EDs in combination with alcohol consumption and sleep deprivation.
  Interventions: Dietary Supplement: Energy Drink, Taurine, Caffeine
- Exercise after consumption (Experimental): Examination of the effects of EDs in combination with alcohol consumption and exercise.
  Interventions: Dietary Supplement: Energy Drink, Taurine, Caffeine

INTERVENTIONS:
Dietary Supplement: Energy Drink, Taurine, Caffeine

SUMMARY:
The aim of this study is to examine the safety and the effects of EDs at high doses, either alone or in combination with other risk factors such as alcohol intake, physical exercise and sleep deprivation, on cardiovascular markers and subjective health.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* healthy (no acute or chronic desease)
* BMI 20,0 - 25,9 kg/m2
* moderate and non-regular consumption of alcohol, EDs and coffee

Exclusion Criteria:

* pregnancy
* regular medication (oral contraceptives permitted)
* hypertension and other deseases of the cardiovascular system
* liver-deseases
* psychiatric deseases
* epilepsy
* other relevant deseases
* (former) alcoholics
* non-compliance to the study-protocol
* simultaneous participation in another clinical trial
* retraction of the written informed consent

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Heart-rate-variability (HRV) | during 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hohenheim, Stuttgart, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Basrai M, Schweinlin A, Menzel J, Mielke H, Weikert C, Dusemund B, Putze K, Watzl B, Lampen A, Bischoff SC. Energy Drinks Induce Acute Cardiovascular and Metabolic Changes Pointing to Potential Risks for Young Adults: A Randomized Controlled Trial. J Nutr. 2019 Mar 1;149(3):441-450. doi: 10.1093/jn/nxy303. PMID 30805607